CLINICAL TRIAL: NCT06091410
Title: Immunogenicity of Concomitant Administration of Omicron-containing COVID-19 Vaccines With Influenza Vaccines : In-depth Immunogenicity Analysis.
Brief Title: Immunogenicity of Concomitant Administration of COVID-19 Vaccines With Influenza Vaccines
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic Kwandong University (Other)
Collaborators: Korea University Guro Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IS23OIME0055
Record Dates: First submitted 2023-10-17; First posted 2023-10-19 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Influenza; Vaccine Reaction; Contaminant Injected
Keywords: COVID-19 vaccine; influenza vaccine; immunogenicity; co-administration
MeSH Terms: conditions — COVID-19; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: prospective, randomized clinical cohort study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- C group (Experimental): concomitant administration of COVID-19 booster and quadrivalent influenza vaccination
  Interventions: Biological: Omicron-containing COVID-19 vaccine; Biological: influenza vaccine
- S group (COVID-19 vaccine only) (Placebo Comparator): separate administration of influenza vaccination followed by COVID-19 booster 4 weeks later
  Interventions: Biological: Omicron-containing COVID-19 vaccine
- S group (influenza vaccine only) (Placebo Comparator): separate administration of influenza vaccination followed by COVID-19 booster 4 weeks later
  Interventions: Biological: influenza vaccine

INTERVENTIONS:
Biological: Omicron-containing COVID-19 vaccine — The COVID-19 vaccine approved for use in the 2023-2024 season
  Arms: C group; S group (COVID-19 vaccine only)
Biological: influenza vaccine — inactivated vaccine containing 15μg hemagglutinin antigen/strain in each 0.5-mL dose, containing four influenza vaccine strains from the 2023-2024 northern hemisphere season
  Arms: C group; S group (influenza vaccine only)

SUMMARY:
The goal is to evaluate the in-depth immunogenicity analysis (including B-cell and T-cell response) of coadministration of a omicron-containing COVID-19 vaccine and influenza vaccine among healthy adults during 2023-24 season.

DETAILED DESCRIPTION:
This was an open-label, randomized clinical trial conducted at the International St. Mary's Hospital in Incheon, South Korea. This study included two study groups: Concomitant administration of omicron containing messenger ribonucleic acid (mRNA) COVID-19 booster and quadrivalent influenza vaccination (QIV) and separate administration of influenza vaccination followed by mRNA booster ≥4 weeks later

* immunogenicity analysis : Blood was drawn at baseline and follow-up visit 4 weeks, 3 months, 6 months, 10-12 months after immunization(For the COVID-19 vaccine, additional blood sampling will be conducted one week after vaccination).
* safety analysis : At 7 days after each vaccine dose, the participants were requested to record the occurrence, severity of solicited adverse events (AEs) through a standardized electronic questionnaire. Participants were also asked to record any unsolicited AEs during the 28 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* who agreed to receive both booster COVID-19 vaccine and influenza vaccine
* individuals who have received the COVID-19 vaccine three or more times and have passed at least 3 months after the last vaccination
* individuals with a history of a single SARS-CoV-2 infection during the Omicron outbreak period (January 2022-February 2023)

Exclusion Criteria:

* individuals with a contraindication to any of the vaccine compounds
* individuals with a history of influenza infection within the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
geometric mean titer against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) | at 7, 28 days, 3, 6, and 10-12 months after COVID-19 vaccination
  geometric mean titer against SARS-CoV-2 (Anti-S immunoglobulin G, Neutralizing antibody)

SECONDARY OUTCOMES:
geometric mean titer against four influenza strain | at 28 days and 7 months after influenza vaccination
  geometric mean titer against four influenza strain
vaccine-induced B-cell responses | at 7, 28 days, 6, and 10-12 months after COVID-19 vaccination
  vaccine-induced B-cell responses and their immune interactions between COVID-19 and influenza vaccines
vaccine-induced CD4+ T cell responses | at 7, 28 days, 6, and 10-12 months after COVID-19 vaccination
  vaccine-induced CD4+ T cell responses and their immune interactions between COVID-19 and influenza vaccines
The incidence rate of adverse events | within 28 days
  The incidence rate of adverse events within 7 days, 28 days, and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Min Joo Choi, Principal Investigator — International St. Mary's Hospital
Locations (2):
- South Korea (2):
  - Korea University Guro Hospital, Seoul, Guro-gu
  - International St. Mary's hospital, Incheon, Seo-gu

IPD SHARING:
Plan to Share IPD: No